CLINICAL TRIAL: NCT05846893
Title: Randomised Trial of Drug-Coated Balloon Versus Drug-Eluting Stent for Clinical Outcomes in Patients With Large Coronary Artery Disease
Brief Title: Drug-Coated Balloon vs. Drug-Eluting Stent for Clinical Outcomes in Patients With Large Coronary Artery Disease
Acronym: REVERSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Medical Industries Sdn. Bhd. (Industry)
Collaborators: B. Braun Melsungen AG (Industry); Ulsan University Hospital (Other); European Cardiovascular Research Center (Network); Seoul National University Hospital (Other); Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-2124
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Coronary Stenosis; De Novo Stenosis
Keywords: de novo; large vessel; coronary artery disease; cardiovascular disease; coronary occlusion; heart disease; acute coronary syndrome; angina; ischemia; stenosis; percutaneous coronary intervention; angioplasty; drug-coated balloon; drug-eluting stent; SeQuent Please; randomised trial
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Coronary Stenosis; Cardiovascular Diseases; Coronary Occlusion; Heart Diseases; Angina Pectoris; Ischemia; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SeQuent® Please NEO drug-coated balloon catheter (Experimental)
  Interventions: Device: SeQuent® Please NEO drug-coated balloon catheter
- Current-generation drug-eluting stent (Experimental)
  Interventions: Device: Current-generation drug-eluting stent

INTERVENTIONS:
Device: SeQuent® Please NEO drug-coated balloon catheter — Treatment of coronary artery disease with SeQuent® Please NEO for de novo lesions in native large coronary arteries
  Arms: SeQuent® Please NEO drug-coated balloon catheter
Device: Current-generation drug-eluting stent — Treatment of coronary artery disease with current-generation drug-eluting stent for de novo lesions in native large coronary arteries
  Arms: Current-generation drug-eluting stent

SUMMARY:
Prospective, randomised, open-label, international multicenter trial to evaluate the safety and efficacy of drug-coated balloon (DCB) treatment compared to drug-eluting stenting (DES) in patients with large coronary artery disease.

DETAILED DESCRIPTION:
Although several reports suggested that DCB application was safe for larger coronary artery lesions and showed good long-term outcomes, there is limited randomised controlled trial (RCT) data on the safety and efficacy of DCB in large coronary artery disease.

Therefore, the study aims to demonstrate the non-inferiority of the drug-coated balloon (DCB) treatment against current-generation drug-eluting stenting (DES) in patients with de novo lesions in large coronary artery disease (reference vessel diameter ≥3.0 mm by visual estimation).

The hypothesis of the study is the clinical outcomes of patients treated with DCB are non-inferior to those treated with current-generation DES.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related:

  1. Patient must be ≥ 18 years of age
  2. Patient is able to verbally confirm understanding of the study aim, risks, benefits, and treatment alternatives of receiving DCB or DES and he/she or his/her legally authorized representative provides written informed consent prior to any study-related procedure
  3. (i) Clinical evidence of angina, and/or (ii) an abnormal functional study demonstrating myocardial ischemia due to the target lesion(s), or (iii) acute coronary syndrome [unstable angina or non-ST-elevation myocardial infarction (NSTEMI) or uneventful STEMI (≥ 48 hours after primary PCI and no sign of thrombus in lesion(s) to treat)]
  4. Patient with lesions suitable for PCI with a DCB (and/or DES) according to the Instructions for Use
  5. Patient is able to comply with the study protocol and agrees to undergo the clinical follow-up of 30 days, 6 months, 12 months, 24 months, and 36 months
* Lesion-related:

  1. Presence of significant de novo large vessel coronary artery disease (reference vessel diameter ≥3.0 mm by visual estimation) with either ≥ 70% diameter stenosis or intermediate ≥ 50% to <70% diameter stenosis with abnormal functional test or symptom of ischemia
  2. Successful lesion preparation. For randomisation, the lesion must satisfy the following criteria after optimal balloon angioplasty: no flow-limiting dissection (TIMI=3), and residual stenosis is ≤ 30%
* Multivessel disease with two or more vessels showing diameter stenosis of 50% or more is not an exclusion as long as it fulfills all study's eligibility criteria.
* In diffuse lesion, inclusion is possible if the proximal reference vessel diameter is 3.0 mm or more.

Exclusion Criteria:

* Patient-related:

  1. Intolerance or allergy to Paclitaxel and/or the delivery matrix (main ingredient: Iopromide)
  2. Severe allergy to contrast media
  3. Recent STEMI (ongoing or < 48 hours after primary PCI and/or has sign of thrombus in lesion(s) to treat)
  4. NSTEMI hemodynamically unstable
  5. Known left ventricular ejection fraction of <30%
  6. Inability to take dual antiplatelet therapy or anticoagulation, or single antiplatelet therapy for at least six months
  7. Non-cardiac co-morbid conditions that may result in protocol non-compliance and inability of patient to complete the study (per the site investigator's medical judgment)
  8. Patient with concomitant medical illnesses that require cytostatic, radiation therapy or renal replacement therapy
  9. Patient who is currently/ planning to participate in another clinical trial when such participation could confound the treatment or outcomes of this study, except for observational registry
  10. Pregnancy or lactation
  11. Patient under administrative or judicial custody
* Lesion-related:

  1. Small vessel disease, defined as <3.0 mm of reference vessel diameter by visual estimation
  2. In-stent restenosis lesions for study lesions
  3. Patient will be excluded if meet any of the following angiographic exclusion criteria after lesion preparation:

     (i) Flow limiting dissection with TIMI flow < III (ii) Residual diameter stenosis >30%

     * The case of persistent ischemic symptoms/signs is up to the operator's decision
  4. Lesions which are untreatable with PCI or other interventional techniques and coronary artery spasm in the absence of a significant stenosis
  5. Left main disease or aorta-ostial lesion requiring revascularization
  6. Severely calcified or tortuous vessels precluding DCB or DES application
  7. Prior Coronary Artery Bypass Graft (CABG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1436 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical Event (NACE) | At 1 year
  Net adverse clinical event (NACE): a composite of all-cause death, non-fatal myocardial infarction, clinically driven target vessel revascularization, or major bleeding (BARC type 3 to 5)

SECONDARY OUTCOMES:
All-cause death | At 12, 24, and 36 months
Non-fatal myocardial infarction | At 12, 24, and 36 months
Clinically driven target vessel revascularization | At 12, 24, and 36 months
Major bleeding (BARC type 3 to 5) | At 12, 24, and 36 months
Cardiac death | At 12, 24, and 36 months
Target vessel myocardial infarction | At 12, 24, and 36 months
Periprocedural myocardial infarction | At 12, 24, and 36 months
Target lesion revascularization | At 12, 24, and 36 months
Stent/lesion thrombosis in treated lesion defined according to the Academic Research Consortium-2 (ARC-2) criteria | At 12, 24, and 36 months
Rehospitalization related to study endpoints | At 30 days, 12 months, 24 months, and 36 months
  Rate of hospitalization related to study endpoints
Stroke (ischemic and hemorrhagic) | At 12, 24, and 36 months
  Number of participants with stroke (ischemic and hemorrhagic)
Total angioplasty procedure time | During the index procedure
Fluoroscopy time of the angioplasty procedure | During the index procedure
Contrast volume of the angioplasty procedure | During the index procedure
Number of devices (DCB/ DES) used for PCI treatment | During the index procedure

OTHER OUTCOMES:
Late lumen loss (LLL) | At 9-12 months post-procedure
  LLL is defined as: the minimal lumen diameter (MLD) immediately after PCI minus the MLD at the follow-up.
Percentage of diameter stenosis | At 9-12 months post-procedure
Minimal lumen diameter | At 9-12 months post-procedure
Binary restenosis | At 9-12 months post-procedure
Quality of life analysis | After 12, 24, and 36 months
  Quality of life analysis using EQ-5D-5L questionnaire
Incidence of angina | At baseline and 12 months
Dual Antiplatelet Therapy (DAPT) duration | At 30 days, 6 months, and 12 months
Comparison of NACE between DCB vs. DES in sex difference, diabetes mellitus, and multivessel disease patients | At 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Seok Shin, MD, Ph.D, Study Chair — Ulsan University Hospital
Locations (19):
- Malaysia (6):
  - Queen Elizabeth II Hospital, Kota Kinabalu, Sabah
  - Sarawak Heart Center, Kuching, Sarawak
  - Sultan Idris Shah Serdang Hospital, Kajang, Selangor
  - National Heart Institute Malaysia, Kuala Lumpur
  - Cardiac Vascular Sentral Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Singapore (3):
  - Tan Tock Seng Hospital, Novena
  - National Heart Centre Singapore, Singapore
  - Khoo Teck Puat Hospital, Singapore
- South Korea (7):
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Gyeongsang National University Changwon Hospital, Changwon, Gyeongsangnam-do
  - Ulsan University Hospital, Donggu, Ulsan
  - Keimyung University Dongsan Hospital, Daegu
  - Kangbuk Samsung Hospital, Seoul
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No